CLINICAL TRIAL: NCT05712928
Title: The Effects of Telehealth Dance/Movement Therapy on People With Chronic Schizophrenia
Brief Title: eMove - Dance/Movement Therapy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2104008484
Record Dates: First submitted 2022-03-14; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Dance/movement therapy; Creative arts therapies; Telehealth dance/movement therapy; Non-pharmacological intervention; Online intervention; Psychosocial functioning
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dance/movement therapy (Experimental): Ten weekly 60-minute individual dance/movement therapy telehealth sessions (eMove).
  Interventions: Behavioral: Dance/movement therapy (eMove)

INTERVENTIONS:
Behavioral: Dance/movement therapy (eMove) — Ten weekly 60-minute individual dance/movement therapy telehealth sessions (eMove) delivered by a board-certified dance/movement therapist. eMove treatment protocol integrates movement techniques, creative embodiment, the non-verbal aspects of self-awareness and interpersonal communication in treatment. eMove sessions focus on helping the participant to increase physical activity level, increasing participants' energy levels and motivation to stay active and better cope with everyday activities, improving overall functioning; reducing severity of negative symptoms of schizophrenia; and providing participants with a sense of connection and social support by connecting with a therapist. In addition, sessions are individualized to the participant's presenting needs.

SUMMARY:
Schizophrenia is a chronic and severe mental disorder affecting 20 million people throughout the world and is the fourth leading cause of disability in the developed world. Currently, restrictions due to the COVID-19 pandemic, cause greater social withdrawal, reduced access to social support, lack of motivation, under-activity and loneliness for patients with schizophrenia. Given the prevalence of under-activity, interventions such as dance/movement therapy that use movement and dance to support intellectual, emotional, and motor functions of the body, can optimize the functioning of individuals with schizophrenia. There have been urgent calls for research on telehealth interventions to address the mental health needs caused by COVID-19 pandemic. To address this call, this study will test the feasibility and acceptability of a novel, 10-week dance/movement therapy protocol to promote activation in chronic schizophrenia designed for telehealth delivery. This study will be the first to examine the feasibility and preliminary effects of telehealth dance/movement therapy to promote activation in chronic schizophrenia. This study can contribute towards the development of telehealth interventions for treatment and rehabilitation of individuals with chronic schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a chronic and severe mental disorder affecting 20 million people throughout the world and is the fourth leading cause of disability in the developed world. Anhedonia, apathy, social withdrawal, and under-activity are common negative symptoms that have a detrimental impact on patients' overall quality of life. Activation, defined as physical, psychological and social engagement in everyday activities, is one of the most important psychosocial predictors of functional outcomes in people with schizophrenia. Psychosocial interventions designed to decrease negative symptoms and improve activation are considered crucial in the treatment of schizophrenia. Movement/body based interventions are one type of psychosocial interventions that are recommended. Given the prevalence of under-activity, interventions such as dance/movement therapy that focuses on movement behavior, emotional expression and social support, can optimize the functioning of individuals with schizophrenia. In addition, as many people with schizophrenia are treated on an outpatient basis and rarely require hospitalization, COVID-19 restrictions cause greater social withdrawal, reduced access to social support, lack of motivation, under-activity, and loneliness. Dance/movement therapy as a therapeutic holistic approach has unique potential to promote activity engagement in individuals with schizophrenia. Preliminary evidence suggests that dance/movement therapy enhances psychosocial functioning and reduces severity of negative symptoms of schizophrenia however to date no study has examined a telehealth delivery of dance/movement therapy to promote activation in this population. Therefore, the overarching goals of this feasibility study are (1) to evaluate the feasibility, acceptability and credibility of a telehealth dance/movement therapy treatment procedures and research protocol; (2) to assess and improve methodological procedures for conducting a randomized controlled trial (RCT) test of telehealth dance/movement therapy protocol; and (3) to determine preliminary effects of telehealth dance/movement therapy to promote activation in chronic schizophrenia. This feasibility study uses a single-group convergent mixed methods design in which quantitative (survey data) and qualitative (semi-structured exit interviews) data are collected concurrently and analyzed independently; the results are then compared and contrasted. The quantitative strand of the study will be a one-group pre/post-test design. For the qualitative strand, we will conduct semi-structured exit interviews post-intervention. The qualitative data will help to (1) obtain participant feedback on the intervention and its telehealth delivery, and (2) enhance our understanding of the impact of the intervention on activation in chronic schizophrenia.

This is the first study to examine the feasibility and preliminary effects of telehealth dance/movement therapy to promote activation in chronic schizophrenia. The findings from this study will provide (1) important methodological and protocol data and substantive pilot data necessary for the next phase of this line of research (a fully powered RCT to evaluate efficacy of treatment); and (2) will contribute towards the development of telehealth interventions for treatment and rehabilitation of individuals with chronic schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Schizophrenia or schizoaffective disorder diagnosis,
* Able to speak and write English,
* Able to attend sessions via Zoom (including internet connection and a device with camera).

Exclusion Criteria:

* An organic brain disease or substance abuse as the primary diagnosis,
* A diagnosis of dementia or cognitive impairment that would interfere with competence to consent to participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Recruitment rates | Baseline
  Proportion of participants enrolled relative to total trial referrals
Consent rates | Baseline
  Proportion of participants consented relative to total trial referrals
Attrition rates | 12 weeks following receipt of treatment
  Proportion of participants who dropped-out/withdrawn relative to total enrolled including reason for drop-out/withdrawal
Treatment compliance | 12 weeks following receipt of treatment
  Number of participants who completed 10 eMove sessions
Treatment acceptance | 12 weeks
  Exit interview based on an interview protocol developed by the researcher
Measurement completion | 12 weeks following receipt of treatment
  Proportion of participants who complete questionnaires
Measurement burden | Through study completion, a maximum of 12 weeks
  Ease to understand, quantity of questions, and fatigued experienced while completing the outcome assessments will be assessed during exit interview
Treatment Fidelity | Through study completion, a maximum of 12 weeks
  Treatment fidelity questionnaire developed by the researcher; (range: 1 to 25 items; A total score of 80% and higher reflects adequate treatment fidelity).
Negative Symptoms (Self-report) | Change from Baseline Psychosocial Illness Impact at post-treatment (week 12) time point
  Measured by Self-evaluation of Negative Symptoms (SNS), a self-assessment of 20 items, allowing patients to evaluate themselves on the five dimensions of negative symptoms: social withdrawal, emotional range, alogia, avolition, and anhedonia. Each item is scored as either 2 (strongly agree), 1 (somewhat agree), or 0 (strongly disagree). The total score is the sum of the 20 items, ranging from 0 (no negative symptoms) to 40 (severe negative symptoms).
Negative Symptoms (Clinical assessment) | Change from Baseline Psychosocial Illness Impact at post-treatment (week 12) time point
  Measured by Brief Negative Symptom Scale (BNSS) is a 13-item instrument, organized into 6 subscales, that asses negative symptoms (anhedonia, distress, asociality, avolition, blunted affect, and alogia). Items are scored on a 0 to 6 scale, with 0 indicating the symptom is absent and 6 indicating the symptom is severe. Items are summed for a total score that ranges between 0 and 78. The BNSS is administered as a semi-structured interview.
Functional impairment (Self-report) | Change from Baseline Psychosocial Illness Impact at post-treatment (week 12) time point
  Measured by Sheehan Disability Scale (SDS), a 3 items self-report questionnaire assessing the extent that symptoms have caused the functional impairment in three inter-related domains; work/school, social and family life. The 3 items are measured on a 10 point visual analog scale. A single score of 5 or greater on any of the three scales are associated with significant functional impairment. The 3 items can also be summed into a single dimensional measure of global functional impairment that rages from 0 (unimpaired) to 30 (highly impaired).
Health and disability (Self-report) | Change from Baseline Psychosocial Illness Impact at post-treatment (week 12) time point
  Measured by World Health Organization - Disability Assessment Schedule (WHODAS) 2.0 a 36-item self-report questionnaire assessing health and disability across six domains: cognition, mobility, self-care, getting along, life activities and participation. The 36 items are rated on a five-point Likert scale. The total score ranges from 0 to 100, higher scores representing greater disability.
Movement assessment (Clinical assessment) | Through study completion, a maximum of 12 weeks
  Measured by Movement Psychodiagnostic Inventory's (MPI) Action Inventory for Movement Session, an 15-item inventory measuring participation, self-related actions, eye contact, orientation, movement changes, types of interaction, torso/limb configurations while moving. (range: 0-2; higher scores reflect less action (higher severity in movement))

SECONDARY OUTCOMES:
Patient Perception of Change (Self-report) | post-treatment, week 12 time point
  Measured by Patient's Global Impression of Change (PGIC) scale, a single item self-report scale (range: 1 (No change) to 7 (a great deal better)).
Psychosocial Illness Impact (Self-report) | Change from Baseline Psychosocial Illness Impact at post-treatment (week 12) time point
  Measured by PROMIS® Psychosocial Illness Impact - Negative - Scale, a 5-point (from 1= Not at all to 5= Very much) rating scale is used in each of the 8 items; higher results mean more severe illness impact on functioning.
Affect (Self-report) | Change from Baseline Psychosocial Illness Impact at post-treatment (week 12) time point
  Measured by PROMIS® Positive Affect Scale, A 5-point (from 1= Not at all to 5= Very much) rating scale is used in each of the 7 items; higher results mean better positive affect.
Clinical Global Impression - Severity of Illness (Clinical assessment) | Change from Baseline Psychosocial Illness Impact at post-treatment (week 12) time point
  Measured by Clinical Global Impression (Severity of Illness [CGI-S]) is a single item 7-point scale measure of severity of illness. Range of responses from 1 (normal) through to 7 (amongst the most severely ill patients).
Clinical Global Impression - Global Improvement (Clinical assessment) | Change from Baseline Psychosocial Illness Impact at post-treatment (week 12) time point
  Measured by Clinical Global Impression (Measured by Global Improvement [CGI-I]) is a single item 7-point scale measure of global improvement. Range of responses from 1 (very much improved) through to 7 (very much worse).

CONTACTS AND LOCATIONS:
Overall Officials: Joke Bradt, PhD, Principal Investigator — Drexel University; Karolina Bryl, PhD, Principal Investigator — Drexel Unviersity
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No